CLINICAL TRIAL: NCT01367236
Title: A Randomised, Prospective Study, Assessing Changes in Cerebral Function in Treatment Naive HIV-1 Infected Subjects Commencing Either Boosted Atazanavir With Truvada or Boosted Darunavir With Maraviroc and Kivexa.
Brief Title: Changes in Cerebral Function in Treatment Naive HIV-1 Infected Subjects Commencing Either Boosted Atazanavir With Truvada or Boosted Darunavir With Maraviroc and Kivexa
Acronym: CogUK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1733; 2011-002656-14 (EudraCT Number)
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: HIV; Impaired Cognition
Keywords: HIV
MeSH Terms: conditions — Cognition Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Active Comparator): treatment with:
  * atazanavir 300 mg daily
  * ritonavir 100 mg daily
  * tenofovir 245 mg daily*
  * emtricitabine 200 mg daily* * as the fixed dose combination Truvada™
  Interventions: Drug: standard care
- Novel therapeutic approach (Active Comparator): * darunavir 800 mg daily
  * ritonavir 100 mg daily
  * lamivudine 300 mg daily**
  * abacavir 600 mg daily**
  * maraviroc 150 mg once daily ** as the fixed dose combination Kivexa ™
  Interventions: Drug: novel treatment

INTERVENTIONS:
Drug: standard care — * atazanavir 300 mg daily
  * ritonavir 100 mg daily
  * tenofovir 245 mg daily*
  * emtricitabine 200 mg daily*
  Arms: standard care
Drug: novel treatment — * darunavir 800 mg daily
  * ritonavir 100 mg daily
  * lamivudine 300 mg daily** and abacavir 600mgs daily**
  * maraviroc 150 mg once daily
  Arms: Novel therapeutic approach

SUMMARY:
The purpose of this study is to compare two different combination anti-HIV therapies over 48 weeks and to assess if differences in improvement in the function of the brain are observed over this period.

The study will compare anti-HIV therapy combinations which are currently in use.

The patients will not have had any previous treatment for their HIV infection.

DETAILED DESCRIPTION:
Impairment in neurocognitive(NC) function in HIV-infected subjects in the current anti-retroviraltreatment (cART) era has been associated with poor compliance with cART, reduced quality-of-life and increased mortality. Reported factors associated with the development of NC function impairment in HIV disease and risks associated with progression of such impairment include degree of immune suppression related to HIV infection, other chronic viral infections (such as chronic hepatitis C co-infection), age and central nervous system (CNS) antiretroviral drug exposure.

One modifiable factor which may be associated with the evolution of NC function impairment is the direct effect of cART on the central-nervous-system (CNS). Certain antiretroviral drugs such as zidovudine, lamivudine, abacavir, nevirapine, efavirenz and indinavir are known to achieve optimal exposure in the cerebro-spinal-fluid (CSF) whereas other drugs, such as the majority of the HIV-1 protease inhibitors penetrate less effectively. Studies to date suggest different cART regimens may have differing effects on NC performance. In the EuroSIDA study, the use of nucleoside-reverse-transcriptase inhibitors was found to specifically protect against the development of HIV related brain disease. More recently, in a small prospective study, ALTAIR, different effect on cerebral function was reported in subjects randomised to commence three different cART regimens.

The investigators propose, in a prospective, randomised study to assess the effects of two different antiretroviral regimens on NC function in HIV infected subjects commencing antiretroviral therapy for the first time.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* signed informed consent
* no previous antiretroviral treatment since HIV diagnosis
* screening CD4+ lymphocyte count <= 350 cells/ųL
* susceptible to all currently licensed (Nucleoside Reverse Transcriptase Inhibitors) NRTIs, (Non-Nucleoside Reverse Transcriptase Inhibitors) NNRTIs and PIs based on HIV-1 genotypic resistance report
* CCR5-tropic HIV based on genotypic resistance testing*

Exclusion Criteria:

* • existing neurological disease

  * hepatitis B or hepatitis C co-infection
  * age under 18 years
  * screening laboratory parameters > grade 2 (with the exception of cholesterol and triglycerides)
  * current history of major depression or psychosis
  * recent head injury (past three months)
  * current alcohol abuse or drug dependence
  * active opportunistic infection or significant co-morbidities
  * patients who are receiving other concomitant medication which are not permitted, as listed in appendix 2
  * female patients of child-bearing potential who:

    * have a positive serum pregnancy test at screening or during the study
    * are breast feeding
    * are planning to become pregnant
  * all participants unwilling to use a barrier method of contraception
  * patients who in the opinion of the investigator are not candidates for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, Principal Investigator — Imperial College London
Locations (6):
- United Kingdom (6):
  - Birmingham Heartlands Hospital:, Birmingham
  - Brighton and Sussex University Hospital NHS Trust:, Brighton
  - Kings College Hospital, London
  - Chelsea and Westminster Hospital NHS Trust, London
  - St. Mary's Hospital, London
  - St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mora-Peris B, Bouliotis G, Ranjababu K, Clarke A, Post FA, Nelson M, Burgess L, Tiraboschi J, Khoo S, Taylor S, Ashby D, Winston A. Changes in cerebral function parameters with maraviroc-intensified antiretroviral therapy in treatment naive HIV-positive individuals. AIDS. 2018 May 15;32(8):1007-1015. doi: 10.1097/QAD.0000000000001786. PMID 29438199

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Boosted: Treatment with:
  tenofovir disoproxil fumarate/emtricitabine 300/200mg atazanavir/ritonavir 300/100mg all once daily
- Maraviroc-intesified Boosted: Treatment with:
  abacavir/lamivudine 600/300mg darunavir/ ritonavir 800/100 mg maraviroc 150mg all once daily
Period: Overall Study
Arm/Group | Standard Boosted | Maraviroc-intesified Boosted
Started | 30 | 30
Completed | 27 | 29
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Boosted | Maraviroc-intesified Boosted | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 31 [27 to 38] | 35 [28 to 41] | 33 [28 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 29 | 29 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 23 | 22 | 45
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 60
Baseline CD4+ cell count [Mean (Standard Deviation); unit: cells/ug] | 453 (218) | 429 (240) | 441 (227)
Baseline HIV RNA [Median (Inter-Quartile Range); unit: copies/ml 10^3] | 45 [22 to 70] | 51 [26 to 76] | 46 [21 to 76]

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function, Global Cognitive Score (Z-score)
Description: When commencing antiretroviral therapy (anti-HIV therapy) for the first time, improvements in the function of the brain are frequently observed. For example memory and concentration may improve. However, whether these improvements may differ between different anti-HIV therapies is largely unknown.
  The purpose of this study is to compare two different combination anti-HIV therapies over 48 weeks and to assess if differences in improvement in the function of the brain are observed over this period.
  Score increase means improved performance of cognitive function
Time Frame: 24 weeks, 48 weeks
Measure: Mean (Standard Error); unit: z score
Arm/Group | Standard Boosted | Maraviroc-intesified Boosted
Number analyzed (Participants) | 27 | 29
z score
  24 weeks | 0.15 (0.07) | 0.19 (0.07)
  48 weeks | 0.16 (0.09) | 0.25 (0.08)
Statistical Analysis 1: Comparison: Standard Boosted vs Maraviroc-intesified Boosted; 24 weeks; Test type: Superiority; p = 0.68, Regression, Linear
Statistical Analysis 2: Comparison: Standard Boosted vs Maraviroc-intesified Boosted; 48 weeks; Test type: Superiority; p = 0.43, Regression, Linear

2. Secondary Outcome: Brain Function, Absolute Change Over 48 Weeks of N-acetyl Aspartate/Creatinine Ratio
Description: The study team will assess the brain functions at each visit. The results of the MRI scans will be compared, changes in N-acetyl aspartate/creatinine ratio over 48 weeks.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ratio of N-acetyl aspartate/creatin
Arm/Group | Standard Boosted | Maraviroc-intesified Boosted
Number analyzed (Participants) | 22 | 26
ratio of N-acetyl aspartate/creatin | 0.071 (0.157) | -0.097 (0.185)
Statistical Analysis 1: Comparison: Standard Boosted vs Maraviroc-intesified Boosted; Test type: Superiority; p = 0.0009, Regression, Linear

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard Boosted | Maraviroc-intesified Boosted
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes